CLINICAL TRIAL: NCT03244059
Title: Proof-of-concept Randomized, Double-blind, Phase IIa Study to Show Feasibility, Validate Assays and Approaches, and Explore Dosing and Safety of Belimumab in Pulmonary Emphysema Patients
Brief Title: Belimumab Treatment of Emphysema Patients With Anti-GRP78 Autoantibodies
Acronym: BOTEGA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Mark Dransfield, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-300000119
Record Dates: First submitted 2017-08-03; First posted 2017-08-09 (Actual); Results first posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Emphysema
Keywords: COPD; belimumab; biologic agent; GRP78
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — belimumab

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to receive active:placebo in a ratio of 2:1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded placebo controlled randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Belimumab (Experimental): Subjects randomized to the experimental treatment arm will receive i.v. administrations of belimumab (10 mg/kg), consisting of three "loading" doses, two weeks apart, followed by five (5) more monthly infusions. The final assessment will be performed at month 8.
  Interventions: Biological: Belimumab
- Placebo (Placebo Comparator): These subjects will be treated with identically appearing placebo i.v. on the same schedule as the experimental arm subjects (i.e., three "loading" doses, two weeks apart, followed by five more monthly infusions. Again, the final assessment will be performed at month 7 (210+10 days after treatment start).
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Belimumab — Belimumab is an anti-BLyS (B-lymphocyte stimulating factor) agent administered by infusion.
  Other Names: Benlysta
  Arms: Belimumab
Drug: Placebo — An identically appearing placebo infusion.
  Arms: Placebo

SUMMARY:
This is intended to be an initial "proof-of-concept" study to show feasibility, validate assays and approaches, and explore dosing and safety of belimumab in pulmonary emphysema patients who have clinically relevant (and quantifiable) autoimmune responses. The primary goal is to determine effects of belimumab on levels of autoantibodies against glucose regulated protein 78 (GRP78) among patients with pulmonary emphysema attributable to cigarette smoking. The investigators hypothesize that belimumab treatment will safely reduce circulating levels of autoantibodies that are associated with emphysema, and comorbidities of this lung disease, including atherosclerosis.

DETAILED DESCRIPTION:
Specific Aim 1: To conduct a double-blind, Phase IIa trial, in which 18 former smokers with pulmonary emphysema (per chest CT scans), and circulating anti-GRP78 autoantibody levels >mean normal values (by ELISA), will be randomized 2:1 to belimumab vs. placebo. Subjects will receive 8 infusions of either belimumab or placebo over a 6 month interval. Plasma anti-GRP78 will be measured pre-treatment, and at 1, 3, 5, and 7 months. The investigators hypothesize belimumab therapy will more effectively reduce anti-GRP78 IgG autoantibodies, the primary endpoint of this trial, compared to placebo.

Specific Aim 2: To determine effects of the belimumab therapy on secondary endpoints (at the times detailed for Aim 1) that include levels of pneumococcal-binding antibodies (by ELISA), circulating B-cell numbers and phenotypes (by flow cytometry), and the rate and severity of adverse events (AE) at any time during treatment. The investigators hypothesize belimumab will have dose-related effects on B-cell numbers and their differentiation, while minimally reducing host defense antibodies, and will also have an acceptable AE profile.

ELIGIBILITY:
Inclusion Criteria:

1. A history of past tobacco smoking (>10 pack years), but quit for >6 months at the time of enrollment. Smoking cessation will be confirmed by serum cotinine assays.
2. Pulmonary emphysema per chest CT scans (F950>5%). About 60% of COPD patients followed in the LHC registry meet these criteria.6 Chest CTs are routine, standard of practice evaluations for patients with COPD, so no new radiographic studies will be necessary for this project.
3. Ability and willingness to give informed consent.
4. Plasma anti-GRP78 binding IgG >mean values in former smokers with no lung disease (standardized OD >0.390) (hence this is a "personalized medicine" approach). Of the 330 emphysema subjects assayed for anti-GRP78 to date, 111 (67%) met this criterion.
5. Age 40-75 y.o. COPD is a disease of older individuals.

Exclusion Criteria:

1. History of prior acute COPD exacerbations or no more than one moderate exacerbation in the last year and no exacerbations four months prior to enrollment. A past history of an acute exacerbation is the single biggest risk for recurrence.36 Exclusion of these higher-risk subjects will minimize drop-outs.
2. Oral steroids or cellular immunosuppressant use (e.g., cyclophosphamide) within 6 months.
3. History or clinical or laboratory evidence of other autoimmune syndromes.
4. Inability or unwillingness to complete the treatment and surveillance protocols.
5. Eligible for lung transplant at time of enrollment. This exclusion will mitigate any potential, however slight, that a patient could be rejected for transplantation due to surgeon concerns about this novel therapy (and will also obviate early drop-outs due to transplantation).
6. History of malignant neoplasm within the last 5 years.
7. Evidence of serious suicide risk including any history of suicidal behavior in the last 6 months and/or any suicidal ideation in the last 2 months or those, in the investigator's judgment, pose a significant suicide risk.
8. History of a primary immunodeficiency.
9. Significant IgG deficiency (IgG level < 400 mg/dL).
10. Have an IgA deficiency (IgA level < 10 mg/dL).
11. Currently on any suppressive therapy for a chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster or atypical mycobacteria).
12. Hospitalization for treatment of infection within 60 days of Day 0.
13. Use of parenteral (IV or IM) antibiotics (antibacterials, antivirals, anti-fungals, or anti parasitic agents) within 60 days of Day 0.
14. Current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 365 days prior to Day 0.
15. History of a positive HIV test or positive screening test for HIV.
16. Serologic evidence of current or past Hepatitis B (HB) or Hepatitis C (HC) infection based on positive tests for HBsAg or HBcAb, or HCAb.
17. History of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies.
18. Any other clinically significant abnormal laboratory value in the opinion of the investigator.
19. Any intercurrent significant medical or psychiatric illness that the investigator considers would make the candidate unsuitable for the study.
20. Women of Child Bearing Potential (WCBP) must have a negative serum pregnancy test (either blood or urine) at screening, and agree to 1 of the following:

    Complete abstinence from intercourse from 2 weeks prior to administration of the 1st dose of study agent until 16 weeks after the last dose of study agent (Sexual inactivity by abstinence must be consistent with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception)

    OR

    Consistent and correct use of 1 of the following acceptable methods of birth control for 1 month prior to the start of the study agent, during the study, and 16 weeks after the last dose of study agent:
    * Oral contraceptive, either combined or progestogen alone
    * Injectable progestogen
    * Implants of levonorgestrel or etonogestrel
    * Estrogenic vaginal ring
    * Percutaneous contraceptive patches
    * Intrauterine device (IUD) or intrauterine system (IUS) with <1% failure rate as stated in the product label
    * Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject. For this definition, "documented" refers to the outcome of the investigator's/designee's medical examination of the subject or review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records
    * Double barrier method: condom and occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam/gel/film/cream/suppository)
21. Use of Excluded Medications:

    * Anti-B-cell therapy:

      * Wash out of 5 therapeutic half lives after prior B-cell therapy, or until pharmacodynamic effect would be minimal (e.g., 1 year following rituximab)
    * 365 days Prior to Belimumab:

      * Any biologic investigational agent (e.g., abetimus sodium, anti CD40L antibody, BG9588/ IDEC 131)
    * Investigational agent applies to any drug not approved for sale in the country in which it is being used
    * 30 Days Prior to Belimumab (or 5 half lives, whichever is greater)

      * Any non-biologic investigational agent
    * Investigational agent applies to any drug not approved for sale in the country in which it is being use
    * Live vaccines within 30 days prior to baseline or concurrently with belimumab

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Lung Health Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Specific Aim 1
Arm/Group | Belimumab | Placebo
Started | 11 | 6
Completed | 10 | 6
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Specific Aim 2
Arm/Group | Belimumab | Placebo
Started | 11 | 6
Completed | 10 | 6
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belimumab | Placebo | Total
Number analyzed (Participants) | 11 | 6 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (6) | 69 (6) | 69 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 9 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of Circulating Anti-GRP78 IgG Levels
Description: Anti-GRP78 IgG is a clinically relevant surrogate biomarker of autoimmunity in pulmonary emphysema patients who have clinically relevant (and quantifiable) autoimmune responses
Time Frame: Plasma concentrations of the anti-GRP78 autoantibodies will be measured pre-treatment and at end of treatment at 210 days (or when subject withdraws)
Population: Measured as Optical Density (OD) at 405 nM of ELISA. OD values are proportional to autoantibody concentration.
Measure: Mean (Standard Error); unit: % change
Arm/Group | Belimumab | Placebo
Number analyzed (Participants) | 10 | 6
% change | -17.0 (5.4) | -2.6 (5.1)

2. Secondary Outcome: Percent Change of Pneumococcal Polysaccharide-binding Antibodies
Description: Treatment effects on concentrations of pneumococcal polysaccharide-binding antibodies by ELISA
Time Frame: Prior to treatment and at end of treatment on day 210 (or the conclusion of treatment if subject withdraws)
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Belimumab | Placebo
Number analyzed (Participants) | 10 | 6
Percent change | -14.1 (9.1) | -5.0 (6.5)

3. Secondary Outcome: Percent Change of Circulating B-cells
Description: Treatment effect on relative percentages of circulating B-cells (CD20+) by flow cytometry
Time Frame: Prior to treatment, and at treatment end on day 210 or when subject participation is terminated
Population: analyzed as % of CD20+ cells among peripheral blood mononuclear cells
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Belimumab | Placebo
Number analyzed (Participants) | 10 | 6
Percent change | -12.2 (4.9) | -5.0 (6.5)

4. Secondary Outcome: Adverse Events
Description: Adverse events will be evaluated according to criteria outlined in the National Cancer Institure (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0.
Time Frame: Study start to completion (7 months)
Measure: Number; unit: Adverse events
Arm/Group | Belimumab | Placebo
Number analyzed (Participants) | 10 | 6
Adverse events | 10 | 4

ADVERSE EVENTS:
Time Frame: 210 days or the end of treatment if withdrawn prior to 7 month completion
Description: Adverse event tabulated and classified based on severity.
Arm/Group | Belimumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 4/10 | 0/6
Other Adverse Events (participants affected / at risk) | 4/10 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belimumab (N=10) | Placebo (N=6)
SAE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Gastric carcinoma diagnosed soon after start of treatment. Adjudicated as not related to intervention.
SAE (Cardiac disorders) | 2 (2) | 0 (0) — Two patients soon after beginning treatment had cardiac catheterizations
SAE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Acute exacerbation of COPD.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belimumab (N=10) | Placebo (N=6)
Minor self limited (Nervous system disorders) | 3 (4) | 0 (0) — Head aches
Minor self limited (Nervous system disorders) | 1 (1) | 0 (0) — blurred vision
minor adverse event (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Hyperglycemia
minor adverse event (Gastrointestinal disorders) | 1 (1) | 0 (0) — constipation
minor adverse event (Gastrointestinal disorders) | 2 (2) | 0 (0) — nausea
minor adverse event (Nervous system disorders) | 1 (1) | 0 (0) — fatigue, restless, depressed
minor adverse event (Gastrointestinal disorders) | 0 (0) | 1 (1) — Diarrhea
minor adverse event (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — rash (on foot)
minor adverse event (Hepatobiliary disorders) | 0 (0) | 1 (1) — minor elevation of aspartate aminotransferase
minor adverse event (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Anemia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/59/NCT03244059/Prot_SAP_000.pdf